CLINICAL TRIAL: NCT04256486
Title: Family Model Diabetes Self-Management Education in Faith Based Organizations
Acronym: FDSMEFBO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 229034; 1R01MD013852-01 (NIH)
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes
Keywords: Family Model; Marshallese; Pacific Islander; Diabetes Education
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family DSMES (Experimental)
  Interventions: Behavioral: Family Model Diabetes Self-Management Education and Support
- Wait List (Experimental)
  Interventions: Behavioral: Family Model Diabetes Self-Management Education and Support

INTERVENTIONS:
Behavioral: Family Model Diabetes Self-Management Education and Support — Participants assigned to this arm received an intervention that includes culturally-adapted DSME with their participating family members in a faith based organization setting.

SUMMARY:
This study's objective is to conduct a cluster randomized control study that evaluates the effectiveness of F-DSME (Family Model Diabetes Self-Management Education) when delivered in a group setting in Marshallese Faith Based Organizations (FBO). The F-DSME has shown to be effective when delivered in patients' homes, and the proposed research will allow us to determine the F-DSME's effectiveness in a FBO setting.

ELIGIBILITY:
Inclusion Criteria:

* self-reported Marshallese
* 18 years of age or older
* have T2D (defined as having an HbA1c equal to or greater than 6.5)
* have at least one family member willing to take part

Exclusion Criteria:

* has received DSME in the past five years
* has a condition that makes it unlikely that the participant will be able to follow the protocol, such as terminal illness, non-ambulatory, severe mental illness, severely impaired vision or hearing, eating disorder
* plans to move out of the geographic region

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-08-22 (Actual)

PRIMARY OUTCOMES:
Glycemic Control, Measured by Change in Adjusted Mean HbA1c(%) From Baseline at various time points | Baseline, Immediate Post-intervention, 6 Months Post-intervention, 12 Months Post-intervention, 18 Months Post-intervention, 24 Months Post-intervention
  Measured by Change in Adjusted Mean HbA1c(%) From Baseline to Immediate Post-intervention, 6 Months Post-intervention, 12 Months Post-intervention, 18 Months Post-intervention, and 24 Months Post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Pearl McElfish, Phd, MDA, Principal Investigator — University of Arkansas
Locations (1):
- UAMS Institute for Community Health Innovation, Springdale, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-07-18): https://cdn.clinicaltrials.gov/large-docs/86/NCT04256486/ICF_000.pdf